CLINICAL TRIAL: NCT03947320
Title: A Multicenter Phase III Uncontrolled Open-label Trial to Evaluate Safety and Efficacy and Pharmacokinetics of Recombinant Human Coagulation Factor VIII (SCT800) in Previously Treated Paediatric Patients With Severe Haemophilia A.
Brief Title: Safety,Efficacy and Pharmacokinetics Evaluation of SCT800 in Previously Treated Paediatric Patients With Severe Haemophilia A.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SCT800-A303
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recombinant Human Coagulation FVIII (Experimental): Participant receivedSCT800 for prophylaxis with 25 - 50 IU/kg injection once every other day or three times per week for 6 months.
  Interventions: Drug: Recombinant Human Coagulation FVIII

INTERVENTIONS:
Drug: Recombinant Human Coagulation FVIII — Participant received SCT800 for prophylaxis with 25 - 50 IU/kg injection once every other day or three times per week for 6 months.
  Other Names: SCT800

SUMMARY:
This study is a multicenter phase III uncontrolled open-label trial to evaluate the efficacy,safety and pharmacokinetics of SCT800 in regular prophylaxis and perioperative treatment in patients (<12 years old) with severe hemophilia A who have been previously treated with coagulation factor VIII(FVIII) . This study includes two phases: the screening period and prophylaxis period.Prophylaxis with 25 - 50 IU/kg of SCT800 shall be administered once every other day or three times per week starting from Visit 1 and prophylaxis with SCT800 shall continue for 24 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged <12 years ;
* Male severe (central laboratory tested FVIII:C <1%) hemophilia A patients;
* Previously received FVIII treatment (prophylactic or bleeding treatment), have the relevant records and are verified to have accumulated EDs ≥150 days（6≤age<12years old）and EDs >50 days（age <6 years old）;
* The bleeding treatment records of at least 3 months before screening can be obtained;
* Negative FVIII inhibitor assay results (laboratory tested Nijmegen-Bethesda assay result <0.6 BU/mL);
* HIV negative; if HIV positive, the viral load <200 particles/uL or <400,000 copies/mL, and HIV patients must satisfy CD4+ count >200/μL;
* The patient or his guardian voluntarily signed the Informed Consent Form.

Exclusion Criteria:

* Known allergy to any coagulation factor VIII or any excipient; known allergy to bovine, rodent or hamster bovine;
* Has a history or family history of blood coagulation factor VIII inhibitor;
* Platelet count <100 × 109/L;
* Clinical liver function test ((glutamic-pyruvic transaminase, glutamic-pyruvic transaminase) ≥ five times the upper limit of normal (ULN) or clinical kidney function test （creatinine) ≥ two times the ULN;
* International normalized ratio (INR) >1.5;
* Patients with other coagulation dysfunction diseases in addition to hemophilia A;
* Patients who used any anticoagulant or anti-platelet treatment (including non-steroidal anti-inflammatory drugs [NSAIDs]) within 1 weeks before the first drug administration or who regularly (e.g., daily, every other day) use anticoagulant or anti-platelet treatment within the clinical trial period;
* Patients who used immunomodulator(e.g., immunoglobulin, corticosteroids,alpha-interferon, prednisone [>10 mg/day and >7 days], or comparable drugs, other than anti-retroviral chemotherapy) within two weeks before the first administration of the study drug or during the clinical trial period;
* Administration of any cryoprecipitate, whole blood or plasma within 30 days prior to administration of study drug.
* Patients with other clinically significant diseases, alcoholism, drug abuse, mental disorders or intellectual disabilities;
* Patients with other severe or clinical significant diseases verified by the investigator to be unable to benefit from the clinical study;
* Patients who participated in other clinical studies within one month before the first drug administration (except FVIII trials) and patients who participated in other FVIII clinical trials after signing the Informed Consent Form;

Max Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Hemophilia A is a kind of sex chromosome recessive genetic disease and ofter occurs in male.
Enrollment: 70 (Estimated)
Dates: Start 2019-12-20 (Estimated); Primary Completion 2020-09-20 (Estimated); Study Completion 2020-09-20 (Estimated)

PRIMARY OUTCOMES:
Annualized Bleeding Rate | up to 24 weeks
  Annualized Bleeding Rate（ABR） can be calculated using the following formula: Number of bleeding events in efficacy evaluation period/(number of days in treatment period/365.25)

SECONDARY OUTCOMES:
Annualized joint bleeding rate | up to 24 weeks
  Annualized joint bleeding rate（AJBR） can be calculated using the following formula: Number of joint bleeding events during efficacy evaluation period/(number of days in treatment period/365.25).
FVIII incremental in-vivo recovery | Predose within 30 min，15 min±2 min
  Incremental recovery is determined as the peak factor level recorded in the first hour after infusion and is reported as [IU/ml]/[IU/kg]
Bleeding event treatment efficacy | up to 24 weeks
  The investigator shall evaluate the hemostatic effect after the treatment of every bleeding event of subjects based on a four-point scale(excellent, good, moderate, not relieved).
Elimination Half Life | Predose within 30 min，15 min±2 min、1 hour±5 min，10 hours±30 min，24 hours±1hours and 48 hours±2 hours post-dose
  t1/2; Chromogenic Assay
Clearance | Predose within 30 min，15 min±2 min、1 hour±5 min，10 hours±30 min，24 hours±1hours and 48 hours±2 hours post-dose
  CL; Chromogenic Assay

OTHER OUTCOMES:
Incidence of FVIII inhibitors | up tp 24 weeks
  The Nijmegen-Bethesda assay shall be used to monitor the production of FVIII inhibitors during the trial.